CLINICAL TRIAL: NCT06939556
Title: Development of a High-throughput Serological Testing Platform for Mass Screening Purposes of Both Pediatric and Adult Cohorts
Brief Title: High-throughput Serological Testing of Antibodies Platform
Acronym: DEVHISE
Status: Recruiting | Type: Observational
Sponsor: Istituto Zooprofilattico Sperimentale delle Venezie (Other)
Collaborators: European Union (Other); VERDI Consortium (Unknown); University of Padova (Other)
Responsible Party: Principal Investigator, Francesco Bonfante, Head of the Laboratory of Experimental Animal Models at the SCS6 - Experimental Virology, Istituto Zooprofilattico Sperimentale delle Venezie (IZSVe), Istituto Zooprofilattico Sperimentale delle Venezie
Other Study IDs: Nr. CE_IZSVE 10/2024
Record Dates: First submitted 2025-03-25; First posted 2025-04-23 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Diagnostics; Pandemic Response
Keywords: pandemic preparedness; serology; high-throughput; emergent infectious diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- Adult Cohort: 20-65 years of age
- Pediatric Cohort: 2-10 years of age

SUMMARY:
In the case of large emergency serosurveys, innovation in the sampling techniques is an often neglected, but relevant aspect to facilitate the enrolment of subjects in both adult and paediatric populations. Further, neutralization assays are the first line of response immediately after the emergence of a novel virus in the human population. This study aims at developing at IZSVe 384-format high-throughput neutralization assays for emerging and re-emerging respiratory viruses with pandemic potential to increase the preparedness capacity at both regional and national levels. This diagnostic platform will include the validation of Mitra VAMS devices for gathering blood samples for the diagnostic procedure. The platform will be tested and validated using adult subject-matched serum samples collected by venipuncture and finger-prick with volumetric tip microsampling devices (Mitra VAMS). This comparison will focus on the titration of antibodies against endemic viruses like influenza type A (i.e., seasonal influenza strains, like pdmH1N1 or H3N2) and SARS-CoV-2. The same serological assay will be developed to titrate neutralizing antibodies against emerging pathogens like avian influenza viruses of the H3 and H5 subtypes, Zika virus, and MERS-CoV.

DETAILED DESCRIPTION:
Orthomyxoviridae, Flaviviridae, and Coronaviridae are viral families from which a pandemic/epidemic agent is expected to emerge in the coming years. In particular, highly pathogenic avian influenza viruses of the H5N1 subtype and MERS-CoV are respiratory viruses that are known to cause sporadic infections in humans in vast areas of the world where these infections are endemic in animals. These pathogens are on the high-priority list of the World Health Organization given their potential to increase their fitness in humans, their ability to reassort/recombine with other respiratory agents, and the unpredictable potential to gain human-to-human transmission abilities. Zika and other exotic zoonotic flaviviruses like Dengue, Usutu, or Mayaro viruses are not respiratory pathogens, but the rising temperatures associated with climate change are making the European region a more favorable ecological space for the introduction and maintenance of these viruses.

The development of a serological high-throughput platform for mass screening is a fundamental element in increasing preparedness for pandemic scenarios. In the case of large emergency serosurveys, innovation in the sampling techniques is an often neglected but relevant aspect to facilitate the enrolment of subjects in both adult and paediatric populations. Venipuncture is considered the gold standard for sampling blood. Nonetheless, this method includes several important drawbacks: the great volume that is collected (exceeding 1 ml), its invasiveness, the need for a sterile environment as well as specialized personnel to perform it, and the potential risk of exposure to pathogens, which demands a great effort in sample preparation and shipping conditions (affecting costs) (reviewed in Bossi et al. 2024).

As a result, starting in 1963 with dry blood spots (DBSs), blood microsampling methods, that is, the collection of small volumes (≤150 μl) of capillary blood derived usually through a finger prick, have been proposed. Capillary sampling is a standard procedure for neonatal screening testing and diabetic patients, while venipuncture is the standard approach to blood sampling and, in particular, for those oriented to the screening of antibodies against infectious diseases. The finger and heel-prick techniques have been rarely adopted for the titration of neutralizing antibodies due to the limited volume of sera available and the cumbersome laboratory process required to recover antibodies (i.e., puncturing DBSs, eluting the spots overnight, etc.).

Microsampling devices, known as volumetric tip microsampling (VTM), represent a novel approach to sampling and self-sampling. These tools serve the same purpose as the DBS (i.e., filter papers), which has been commonly used for neonatal hematology, but with the advantage of the ease of automation and the standardization of sample volumes. Further, VTM can be particularly beneficial in remote non-specialized centers and domestic settings where venipuncture is not possible and where logistical impediments challenge the storage of samples.

VTM is a method that permits a correct quantification of the sample. Hematocrit, along with other parameters, such as humidity and drying conditions, influence spot size, spot homogeneity, and extraction recovery of analytes in DBS, making it inadequate for procedures that require quantification of analytes (reviewed in Thangavelu et al. 2023). Moreover, filter paper properties, a fundamental component of DBS, can introduce further bias by influencing "the maximum loading capacity, blood spreadability, chromatographic effects, analyte stability and recovery." (reviewed in Thangavelu et al. 2023).

During epidemic emergencies, laboratories rarely meet high-volume requests for the detection and titration of neutralizing antibodies due to technical and logistical constraints. Hence, there is a need to scale up laboratories' capacities to meet such requests. In the case of a hub for serological surveys, scaling up the existing techniques requires developments in the field of automation (i.e., the use of liquid-handling workstations) and the transition from a serological assay based on the standard 96-well plate to a 384-well plate technology. Working with the 384 format not only meets the need for capacity scale-up but also allows for a reduction in the sample's minimal working volume. Such a reduction of the working volumes would be a positive element for increasing the sensitivity of assays carried out on samples collected through VTM (i.e., avoiding elution steps to meet higher working volumes). Moreover, lower volumes of blood imply minimizing the distress associated with lengthy restraints of pediatric patients (i.e., one drop of blood rather than two or three).

There is a limited body of literature on the use of VTM as an alternative to DBS for the collection of capillary blood. VTM has been mainly compared to serum samples obtained by venipuncture regarding the performance of hemato-biochemical and metabolic profiling analyses. Only one study compared the performance of a neutralization assay targeting antibodies against the respiratory syncytial virus (RSV) using samples obtained by either venipuncture or with VTM, finding that VTM was an adequate device to collect and store the blood samples for viral neutralization assays (Terstappen et al., 2023).

Using a lentiviral expression system neutralization assay, Roper and co-authors proved in 2023 that DBS on filter paper delivered similar results to patient-matched sera in assessing the presence of neutralizing antibodies against SARS-CoV-2. Nonetheless, sensitivity issues were observed in connection to blood spot cut-out size variability. In 2021, Sancilio and co-authors relied on a surrogate virus neutralization test (sVNT) that quantified the inhibition of the interaction between SARS-CoV-2 S and human angiotensin-converting enzyme 2 receptor protein and demonstrated that responses in DBS from SARS-CoV-2 PCR positive and negative samples had a concordance correlation of 99% to paired sera.

Among different blood microsampling methods, "the Mitra device, which comprises a plastic sampler attached to a proprietary hydrophilic polymer tip based on Mitra's patented volumetric absorptive microsampling (VAMS®) technology" (Thangavelu et al. 2023) stands out because it allows for higher volumes of blood to be collected than other VTM devices. Mitra devices are compatible with 96-Autoracks and automated liquid-handling systems, making them exceptionally indicated for high-throughput methods. According to Kok and Fillet's review (2018), "[a] cross-laboratory study showed that the VAMS technology enables the collection of an accurate and precise blood volume regardless of the haematocrit." Like other microsampling devices, Mitra VAMS allows for self-sampling and is minimally invasive. However, beyond these advantages, these devices have further ones: compared to most other microsampling devices, one can collect greater blood volumes; and, as noted above, they are exceptionally compatible with high-throughput processes. These traits make them notable candidates for pandemic preparedness and response. Indeed, Mitra VAMS have been used for procedures aiming at detecting and titrating antibodies against SARS-CoV-2 (e.g., Johnson et al. 2022; Whitcombe et al., 2020; Wang et al. 2020; Klumpp-Thomas et al. 2021).

This study aims to develop at IZSVe 384-format high-throughput neutralization assays for emerging and re-emerging respiratory viruses with pandemic potential to increase the preparedness capacity at both regional and national levels. This diagnostic platform will include the validation of Mitra VAMS devices for gathering blood samples for the diagnostic procedure.

Primary objective: Validate the use in the diagnostic practice of microsampling devices (Mitra VAMS) for the detection of neutralizing antibodies for viral infectious diseases of epidemic nature in a real-world scenario for adult and pediatric populations.

Secondary objective: Develop a high-throughput serological platform for the detection of neutralizing antibodies against avian influenza strains associated with pandemic potential (H5N1, H3N8, H9N2, etc), MERS-CoV and Zika virus.

This study will be a cross-sectional study. It will allow us to evaluate the diagnostic performance of the assay in a real-world setting and to identify potential confounding variables. To validate the microsampling device, we will enroll 62 adult and 90 pediatric patients who will be subjected to venipuncture for either routine diagnostic purposes or routine medical examinations by the occupational physician. For this reason, venipuncture procedures should not be considered as an intervention. In this study, the intervention will consist only of capillary sampling with a lancet (i.e., finger prick). This comparison will focus on the titration of antibodies against endemic viruses like influenza type A (i.e., seasonal influenza strains, like pdmH1N1 or H3N2) and SARS-CoV-2. The same serological assay will be developed to titrate neutralising antibodies against emerging pathogens like avian influenza viruses of the H3 and H5 subtypes, Zika virus, and MERS-CoV.

The study is part of the VERDI (SARS-coV2 Variants Evaluation in pRegnancy and paeDIatrics cohorts) project funded by the European Union.

ELIGIBILITY:
Inclusion Criteria:

Adult Cohort - between 20 and 65 years of age Pediatric Cohort - between 2 and 10 years of age Signed consent form by the subject for adults or by caregivers for children

Exclusion Criteria:

1. subjects with an immunocompromised status, such as immunodeficiency disorders or those undergoing immunosuppressant treatments
2. subjects with underlying chronic inflammatory conditions (i.e., autoimmune disorders, chronic gastrointestinal, and rheumatic conditions)
3. subjects who have received immunomodulatory treatment within the past year.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Employees of the IZSVe between the ages of 20 and 65 years Children admitted at the Department of Women's and Children's Health, Padova University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Detection of neutralising antibodies for viral infectious diseases of epidemic nature | From enrollment to detection of the presence or lack thereof of neutralizing antibodies for seasonal influenza virus and/or SARS-CoV-2 (around 2 months).
  Validation of the use in the diagnostic practice of microsampling devices (Mitra VAMS) for the detection of neutralizing antibodies for viral infectious diseases of epidemic nature in a real-world scenario for adult and pediatric populations.

SECONDARY OUTCOMES:
high-throughput serological platform for the detection of potentially pandemic viruses | From enrollment to development of a high-throughput serological platform for the detection of neutralizing antibodies against avian influenza strains associated with pandemic potential (H5N1, H3N8, H9N2, etc), MERS-CoV and Zika virus (around 5 months).
  Development of a high-throughput serological platform for the detection of neutralizing antibodies against avian influenza strains associated with pandemic potential (H5N1, H3N8, H9N2, etc), MERS-CoV and Zika virus.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Zooprofilattico Sperimentale delle Venezie, Padua, Italy
  - Padova University Hospital, Department of Women's and Children's Health, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
Not needed for the objectives of the study.

REFERENCES:
- [Background] Whitcombe AL, McGregor R, Craigie A, James A, Charlewood R, Lorenz N, Dickson JM, Sheen CR, Koch B, Fox-Lewis S, McAuliffe G, Roberts SA, Morpeth SC, Taylor S, Webb RH, Jack S, Upton A, Ussher JE, Moreland NJ. Comprehensive analysis of SARS-CoV-2 antibody dynamics in New Zealand. Clin Transl Immunology. 2021 Mar 14;10(3):e1261. doi: 10.1002/cti2.1261. eCollection 2021. PMID 33747511
- [Background] Wang Y, Sun J, Li X, Zhu A, Guan W, Sun DQ, Gan M, Niu X, Dai J, Zhang L, Zhang Z, Shi Y, Huang S, Mok CKP, Yang Z, Wang Z, Tan W, Li Y, Chen L, Chen R, Peiris M, Zhong N, Zhao J, Huang J, Zhao J. Increased Pathogenicity and Virulence of Middle East Respiratory Syndrome Coronavirus Clade B In Vitro and In Vivo. J Virol. 2020 Jul 16;94(15):e00861-20. doi: 10.1128/JVI.00861-20. Print 2020 Jul 16. PMID 32434886
- [Background] Thangavelu MU, Wouters B, Kindt A, Reiss IKM, Hankemeier T. Blood microsampling technologies: Innovations and applications in 2022. Anal Sci Adv. 2023 May 18;4(5-6):154-180. doi: 10.1002/ansa.202300011. eCollection 2023 Jul. PMID 38716066
- [Background] Terstappen J, Delemarre EM, Versnel A, White JT, Derrien-Colemyn A, Ruckwardt TJ, Bont LJ, Mazur NI. RSV Neutralizing Antibodies in Dried Blood. J Infect Dis. 2024 Jul 25;230(1):e93-e101. doi: 10.1093/infdis/jiad543. PMID 39052716
- [Background] Sancilio AE, D'Aquila RT, McNally EM, Velez MP, Ison MG, Demonbreun AR, McDade TW. A surrogate virus neutralization test to quantify antibody-mediated inhibition of SARS-CoV-2 in finger stick dried blood spot samples. Sci Rep. 2021 Jul 28;11(1):15321. doi: 10.1038/s41598-021-94653-z. PMID 34321523
- [Background] Roper KJ, Thomas J, Albalawi W, Maddocks E, Dobson S, Alshehri A, Barone FG, Baltazar M, Semple MG, Ho A, Turtle L; ISARIC4C Consortium; Paxton WA, Pollakis G. Quantifying neutralising antibody responses against SARS-CoV-2 in dried blood spots (DBS) and paired sera. Sci Rep. 2023 Sep 11;13(1):15014. doi: 10.1038/s41598-023-41928-2. PMID 37697014
- [Background] Kok MGM, Fillet M. Volumetric absorptive microsampling: Current advances and applications. J Pharm Biomed Anal. 2018 Jan 5;147:288-296. doi: 10.1016/j.jpba.2017.07.029. Epub 2017 Jul 27. PMID 28803682
- [Background] Klumpp-Thomas C, Kalish H, Drew M, Hunsberger S, Snead K, Fay MP, Mehalko J, Shunmugavel A, Wall V, Frank P, Denson JP, Hong M, Gulten G, Messing S, Hicks J, Michael S, Gillette W, Hall MD, Memoli MJ, Esposito D, Sadtler K. Standardization of ELISA protocols for serosurveys of the SARS-CoV-2 pandemic using clinical and at-home blood sampling. Nat Commun. 2021 Jan 4;12(1):113. doi: 10.1038/s41467-020-20383-x. PMID 33397956
- [Background] Johnson, Joseph M., Syrena C. Fernandes, Danica L. Wuelfing, Aaron R. Baillargeon, Evan L. MacLure, Soyoon Hwang, Andrew J. Ball, et al. 2022. "Quantifying Post-Vaccination Protective Anti-SARS-CoV-2 IgG Antibodies in Blood and Saliva with a Fully Automated, High Throughput Digital Immunoassay". Preprint. Infectious Diseases (except HIV/AIDS). https://doi.org/10.1101/2022.01.21.22269165
- [Background] Bossi E, Limo E, Pagani L, Monza N, Serrao S, Denti V, Astarita G, Paglia G. Revolutionizing Blood Collection: Innovations, Applications, and the Potential of Microsampling Technologies for Monitoring Metabolites and Lipids. Metabolites. 2024 Jan 11;14(1):46. doi: 10.3390/metabo14010046. PMID 38248849
- See also: This is the website of the umbrella project. — https://verdiproject.org/